CLINICAL TRIAL: NCT01709851
Title: A Single-center, Open, Pilot Trial to Investigate the Performance of the GlucoMen®Day System Using Intravascular and Subcutaneous Microdialysis in Subjects With Type 1 Diabetes
Brief Title: Performance Study to Test the GlucoMen®Day System Using Intravascular and Subcutaneous Microdialysis in Subjects With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Menarini Group (Industry)
Responsible Party: Sponsor
Other Study IDs: GMD_05
Record Dates: First submitted 2012-10-11; First posted 2012-10-18 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Intravascular continuous glucose monitoring; Subcutaneous continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 Diabetes - vMD and sMD: Patients will undergo vascular (vMD) and subcutaneous microdialysis (sMD) using the GMD-system (GlucoMen(R)Day-system)
  Interventions: Device: Vascular and subcutaneous microdialysis using the GMD-system
- Type 1 diabetes - vMD: Patients will undergo vascular microdialysis (vMD) using the GMD-system (GlucoMen(R)Day-system)
  Interventions: Device: Vascular microdialysis using the GMD-system

INTERVENTIONS:
Device: Vascular microdialysis using the GMD-system — Glucose levels will be monitored by means of vascular microdialysis using the GlucoMen(R)Day system
  Groups: Type 1 diabetes - vMD
Device: Vascular and subcutaneous microdialysis using the GMD-system — Glucose levels will be monitored by means of vascular and subcutaneous microdialysis using the GlucoMen(R)Day system
  Groups: Type 1 Diabetes - vMD and sMD

SUMMARY:
Over the last years, a number of systems for continuous subcutaneous glucose monitoring have been marketed and are routinely used in patients with diabetes to obtain more detailed information about 24-hour glucose profiles.

In the hospital, numerous factors influencing glycemic control and possibly leading to glucose excursions out of the desired range exist, e.g. interventions for which the patient has to remain fasting or medications such as corticosteroids or vasopressors. A reliable continuous glucose signal could help to observe levels of glycaemia not only at defined time-points but continuously, making it possible for physicians and nursing staff to better adjust antihyperglycemic therapy and to react before the patient is exposed to severe hypo- or hyperglycaemia.

In the hospital setting, vascular access is granted in the majority of patients and could as well be used as an alternative site for continuous glucose monitoring.

The aim of the present study is to assess accuracy of the glucose data obtained by means of an intravascular microdialysis-based CGM system against venous blood glucose reference measurements.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained after being advised of the nature of the study
* Male or female aged 18 - 75 years (both inclusive)
* Type 1 diabetes treated with multiple daily insulin injection or continuous subcutaneous insulin infusion for 12 months
* Body mass index 20.0 - 29.5 kg/m² (both inclusive)
* HbA1c < 86.0mmol/mol

Exclusion Criteria:

* Female of childbearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods.
* Skin pathology or condition prohibiting needle insertion as judged by the investigator.
* History of bleeding disorder.
* History of heparin-induced thrombocytopenia (HIT)
* Current participation in another clinical study.
* Significant acute or chronic illness that might interfere with subject safety or integrity of results as judged by the investigator.
* Lipodystrophy
* Current treatment with systemic (oral or i.v.) corticosteroids or any anticoagulation medication.
* Blood donation or blood loss of more than 500 mL within 12 weeks prior to the study day.
* Known hypersensitivity to Fondaparinux sodium (Arixtra®).
* Significant history of alcoholism or drug abuse or a positive result in urine drug/alcohol screen.

Study day exclusion criteria:

* Non-fasting (i.e. consumption of food or beverages, other than water, later than 22:00 hours the evening before the visit) except if slight intake of rapidly absorbable carbohydrates has been necessary in order to prevent hypoglycaemia.
* Positive result of alcohol breath test.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with type 1 diabetes
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Point Accuracy of the microdialysis signal | 72 hours
  MARD (mean absolute relative difference), MARE (mean absolute relative error), %Press analysis

SECONDARY OUTCOMES:
Rate accuracy of the microdialysis signal | 72 hours
  R-EGA (rate error grid analysis) and P-EGA (point error grid analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Dept. of Internal Medicine, Endocrinology and Metabolism, Graz, Austria